CLINICAL TRIAL: NCT02864121
Title: Association Between High-risk HPV Genome Integration Detected by Molecular Combing and Cervical Lesions Severity and/or Evolution
Brief Title: Oncogenous HPV DNA Integration (Intégration De l'ADN Des HPV Oncogènes)
Acronym: IDAHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PI15088
Record Dates: First submitted 2016-05-11; First posted 2016-08-11 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Abnormal Cytology
Keywords: High-risk human papillomavirus; Integration of HR-HPV DNA; biomarker of severity; biomarker of evolution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- arm 1 (Experimental): all patients included in IDAHO study
  Interventions: Other: all patients included in IDAHO study

INTERVENTIONS:
Other: all patients included in IDAHO study

SUMMARY:
High-risk human papillomavirus (HR-HPV) are involved in cervical cancer development. Integration of HR-HPV DNA in cellular genomes is considered as a major event in the cervical cancer development. The aim of this study is to validate the integration of the HPV-HR as an appropriate biomarker of the severity of precancerous lesions and progression of cervical lesions towards cervical cancer. HR-HPV integration status will be analyzed by Molecular Combing technology, which allows direct and high-resolution visualization of the integration of high-risk HPV genomes.

ELIGIBILITY:
Inclusion Criteria:

* women aged from 25 to 65 years
* consulting in a gynecological-obstetrical service of one of the investigator center for a colposcopy reflex after an abnormal cytology dating of less than 6 months and more than 1 month
* signature of the informed consent
* affiliated to Social Security

Exclusion Criteria:

* women vaccinated against HPV
* women who received a treatment for a cervical pathology followed by a normal
* women with a known positive HIV test
* women suffering from a chronic pathology that generate immunosuppression
* Women currently treated with immunosuppressors
* Women treated with corticoids currently or dating of less than 6 months
* protected by law
* pregnant

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
presence of high-risk papillomavirus in the analysis of cervical smear | during 36 months after inclusion
integration of genome of high-risk papillomavirus detected in cervical smear according molecular combing | during 36 months after inclusion
presence and severity of cervical lesion according to results of cervical smear, colonoscopy and histological analysis | during 36 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France